CLINICAL TRIAL: NCT01068873
Title: Kaletra and Maraviroc in Antiretroviral Therapy-Naïve Patients - KALMAR Study -Version 1.0 Amendment 2
Brief Title: Kaletra and Maraviroc in Antiretroviral Therapy (ART)-Naive Patients (KALMAR Study)
Acronym: KALMAR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Temple University (Other)
Collaborators: Abbott (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Temple IRB 12848
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: HIV Infections
Keywords: HIV; Protease Inhibitor; CCR5 Co-receptor Antagonist; treatment naive
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Ritonavir; Maraviroc; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label single arm (Experimental): Drug: lopinavir/ritonavir plus maraviroc
  Interventions: Drug: lopinavir/ritonavir plus maraviroc

INTERVENTIONS:
Drug: lopinavir/ritonavir plus maraviroc — Lopinavir/ritonavir 400 mg/100 mg two tablets twice daily with Maraviroc 150 mg one tablet twice daily will be administered for 48 weeks to participants meeting entry criteria.
  Other Names: Lopinavir/ritonavir (Kaletra); Maraviroc (Selzentry); Nucleoside sparing regimen

SUMMARY:
The primary objective of this pilot study is to assess the efficacy of lopinavir/ritonavir (Kaletra, a protease inhibitor, PI) when used in combination with maraviroc (Selzentry, an HIV entry inhibitor) for the treatment of antiretroviral naïve HIV infected patients. Twenty patients will be enrolled and studied for 48 weeks.

DETAILED DESCRIPTION:
As patients with HIV are living longer it is important to explore antiretroviral treatments which may reduce the development of long term complications while preserving future HIV treatment options. This trial explores an antiretroviral treatment regimen which does not include the nucleoside reverse transcriptase inhibitor class which is thought to have long-term toxicity. This is a non-randomized, open label trial in participants meeting entry requirements.

Participants will be evaluated at screening, baseline,and weeks 4, 8, 12, 24, 36, and 48 to include clinical assessments as well as laboratory assessments.

An interim analysis will be performed when all patients have reached the week 24 visit.

ELIGIBILITY:
Inclusion Criteria:

* The patient has signed and dated approved informed consent form.
* There is confirmed laboratory diagnosis of HIV infection (positive ELISA HIV antibody test confirmed by Western blot, p24 antigen assay, quantitative HIV-1 RNA assay, or HIV culture).
* The patient is at least 18 years of age.
* ART-naïve, lopinavir/ritonavir susceptible on genotypic testing, CCR5-tropic virus on Trofile testing (ESTA).
* Negative pregnancy test within 72 hours prior to start of study for women of childbearing potential.
* Females of childbearing potential and males must utilize effective barrier contraception.
* HIV RNA greater than 1,000 copies per mL at entry.
* Liver enzymes (AST, ALT) < 3 times the upper limit of normal.

Exclusion Criteria:

* Patients who are pregnant or breast-feeding.
* Active alcohol or substance abuse sufficient, in the Investigator's opinion that makes compliance to the study protocol unlikely.
* Suspected or active HIV-related opportunistic infection or condition requiring acute therapy within 30 days of entry into the trial.
* Patients on therapy for hepatitis B.
* Patients with hepatitis B surface antigen, or any evidence of active hepatitis B such as positive hepatitis B DNA and/or presence of hepatitis e antigen or e antibody.
* Acute hepatitis B or C within 60 days of entry.
* Patients harboring preexistent co-receptor CXCR4 tropic or dual-or mixed-tropic HIV.
* Patients harboring HIV resistant to lopinavir/ritonavir on genotypic testing.
* The presence of decompensated heart failure, myocardial infarction within 1 year, bypass surgery, severe vascular disease, or active hepatobiliary disease.
* Concomitant use of rifampin, ergot derivatives (i.e. dihydroergotamine, ergotamine), cisapride, lovastatin, simvastatin, triazolam, orally administered midazolam, carbamazepine, phenytoin, St. John's wort, ketoconazole, itraconazole, clarithromycin, telithromycin, amiodarone, bepridil, flecainide, propafenone, quinidine, voriconazole or nefazodone.
* Patients with concomitant diagnosis of malignancy or cancer other than basal cell carcinoma within the past 5 years.
* Concomitant use of investigational agents including the use of any investigational vaccines.
* Any other clinical conditions or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for study, or unable to comply with the dosing requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary van den Berg-Wolf, MD, Principal Investigator — Temple University
Locations (1):
- Temple General Internal Medicine, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Label Single Arm
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Single Arm
Number analyzed (Participants) | 1
Age, Continuous [Median (Full Range); unit: years] | 29 [29 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Assess Proportion of Participants With HIV RNA Levels <50 and < 400 Copies/mL.
Time Frame: week 48
Population: Subject terminated study prior to week 48
Arm/Group | Open Label Single Arm
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With HIV RNA < 50 and <400 Copies/ml.
Time Frame: week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Single Arm
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Assess the Proportion of Participants at Study Termination With VL < 50 Copies/ml.
Time Frame: week 48
Population: Subject terminated study prior to week 48
Arm/Group | Open Label Single Arm
Number analyzed (Participants) | 0

4. Secondary Outcome: Determine the Time to Viral Suppression (VL < 50 Copies/ml).
Time Frame: 48 weeks
Population: Subject terminated study prior to week 48
Arm/Group | Open Label Single Arm
Number analyzed (Participants) | 0

5. Secondary Outcome: Determine the Median Change in VL From Baseline to Week 24, to Week 48 and to Study Termination.
Time Frame: week 24, week 48
Population: Analysis was not performed as only one subject was enrolled
Arm/Group | Open Label Single Arm
Number analyzed (Participants) | 0

6. Secondary Outcome: Assess the Changes in CD4+ T Cell Count.
Time Frame: week 24, 48
Population: Analysis was not performed because only 1 subject was enrolled and terminated study prior to week 48
Arm/Group | Open Label Single Arm
Number analyzed (Participants) | 0

7. Secondary Outcome: Assess Development of HIV Resistance Mutations and in HIV Co-receptor Tropism Changes in Participants Who Develop Virologic Rebound.
Time Frame: week 48
Population: Subject terminated study prior to week 48
Arm/Group | Open Label Single Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Open Label Single Arm
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes